CLINICAL TRIAL: NCT00156585
Title: Prospective Study of Predictive Value of Dynamic Contrast Enhancement Magnetic Resonance Imaging With Gadolinium on the Response of a Cerebral Tumor to a Treatment With Gamma Knife
Brief Title: Predictive Value of Dynamic Contrast Enhancement MRI on a Cerebral Tumor Response to Gamma Knife Treatment
Status: Completed | Type: Observational
Sponsor: Martin Lepage (Other)
Responsible Party: Sponsor-Investigator, Martin Lepage, MD, Université de Sherbrooke
Organization: Université de Sherbrooke (Other)
Other Study IDs: 05-063
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Cerebral Metastases
Keywords: cerebral metastases; dynamic contrast enhanced magnetic resonance imaging; DCE-MRI; gamma knife

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypothesis: the pattern of MRI contrast enhancement after gadolinium injection is different in tumors that respond well to gamma knife.

We are going to acquire sequential T1-weighted images of brain lesions before, during and after injection of Gd-DTPA. This will be repeated before and after a treatment with gamma knife. We will then analyse our results to see if there are common enhancement characteristics between lesions that will respond well to the radiosurgery treatment. Response will be clinically assessed by tumor volume as determined by MRI approximately 4 to 6 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient with intracerebral lesion benign or malignant wich are not concerned by the exclusion criteria

Exclusion Criteria:

* Pancranial radiotherapy
* Residual postop lesion
* Gliomas
* Patients < 18 years old
* Anterior allergic reaction to gadolinium
* Claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: oncology clinic
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2005-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
MRI parameters | Before treatment with the Gamma Knife
  Tumor volume, Ktrans, ve, time at maximum signal enhancement, maximum signal difference, ADC, basal T1 value

CONTACTS AND LOCATIONS:
Overall Officials: Jean Chenard, MD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Faculté de médecine, Université de Sherbrooke, Sherbrooke, Quebec, Canada